CLINICAL TRIAL: NCT04402840
Title: Stellate Ganglion Block (SGB) for COVID-19 Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Ali Rezai, Director, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004963113
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Acute Respiratory Distress Syndrome; COVID-19
Keywords: Acute Respiratory Distress Syndrome; COVID-19; Autonomic Nervous System; Stellate Ganglion
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stellate Ganglion Block (SGB) (Experimental): Clinical Stellate ganglion block
  Interventions: Procedure: Stellate Ganglion Block

INTERVENTIONS:
Procedure: Stellate Ganglion Block — The procedure will be done at the bedside in the ICU without interfering with ongoing treatment.

SUMMARY:
The purpose of this study is to understand if it is safe and useful to perform SGB (Stellate Ganglion Block) in patients who have severe lung injury Acute Respiratory Distress Syndrome (ARDS) due to COVID-19 infection.

DETAILED DESCRIPTION:
Primary Aim:

• To determine safety of stellate ganglion block (SGB) in ARDS

Secondary Aim:

* To determine efficacy of SGB in slowing the progression of ARDS

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 to 80
* Subjects with PCR documented diagnosis of COVID-19 ARDS requiring critical care and transfer to intensive care unit
* Bilateral opacities consistent with pulmonary edema must be present and may be detected on CT or chest radiograph

Exclusion Criteria:

* Subjects with pre-existing cardiac failure
* Hemodynamic Instability
* Subject on Extracorporeal membrane oxygenation (ECMO)
* Anatomical inability to do a stellate block

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse events related to SGB | 3 Months
  Adverse events that can atleast unlikely be attributed to SGB
All Adverse events | 3 Months
  All adverse events related to COVID-19
Death | 3 Months
  Death due to any cause

SECONDARY OUTCOMES:
Assessment of respiratory/ pulmonary function | 3 Months
  Change from baseline clinical respiratory/pulmonary function as assessed by change in PF ratio
Radiographic criteria | 3 Months
  Change from last imaging data obtained prior to SGB procedure
Cardiac function | 3 Months
  Change from baseline clinical cardiac function as assessed by improvement in arrhythmia as measured by standard of care ECG ( rate, rhythm and / or any aberrant electro physiological changes)

CONTACTS AND LOCATIONS:
Overall Officials: Ali R Rezai, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Rockefeller Neuroscience Institute, Morgantown, West Virginia, United States